CLINICAL TRIAL: NCT04176484
Title: Feasibility of Opportunistic Salpingectomy During Non-Gynecologic Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Sponsor
Other Study IDs: 22001
Record Dates: First submitted 2019-11-21; First posted 2019-11-25 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; Opportunistic salpingectomy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survey: Women, 18 years of age or older, who are scheduled for an abdominal procedure after being seen in the General Surgery clinic will be given a handout (attached) by clinic staff during routine pre-op counseling informing them that they may be called and asked to participate in a research survey. Women age 25 and above who are scheduled for an abdominal procedure and were seen in the General Surgery Clinic will be called and asked to complete a 5-10 minute verbal survey prior to their date of surgery. Some additional information will be gleaned from the medical record during the interview. Participation will be voluntary and all data collected will be recorded without any identifiers.
  Interventions: Other: Survey
- Operating Room Feasibility: A list of women 25 or older who are scheduled for an abdominal procedure after being seen in the General Surgery clinic will be generated to include MRN, procedure date, and pocedure type. A medical record review will be undertaken of these women and we will collect information about conditions that would facilitate or hinder the ability to perform a salpingectomy. No patient interaction will occur by the study team and all data will be de-identified at the time of collection.

INTERVENTIONS:
Other: Survey — Women age 25 and above who are scheduled for an abdominal procedure and were seen in the General Surgery Clinic will be called and asked to complete a 5-10 minute verbal survey prior to their date of surgery. Some additional information will be gleaned from the medical record during the interview.
  Groups: Survey

SUMMARY:
It is now felt that the majority of ovarian cancers originate in the fallopian tubes. Opportunistic salpingectomy has been found to decrease ovarian cancer risk by approximately 65%, with additional removal of the ovaries decreasing risk up to 98%. Using data collected under IRB #21841 and a population based statistics model we found that performing opportunistic salpingectomy during non-gynecologic abdominal surgery could decrease the incidence of ovarian cancer by 28-38%.

DETAILED DESCRIPTION:
The purpose of this study is to:

1. gauge patient interest and
2. evaluate the feasibility of offering opportunistic salpingectomy or salpingo-oophorectomy to women undergoing non-gynecologic surgery at UVA medical center.

Data for this study will be collected in two different ways:

Part 1: Women, 18 years of age or older, who are scheduled for an abdominal procedure after being seen in the General Surgery clinic will be given a handout (attached) by clinic staff during routine pre-op counseling informing them that they may be called and asked to participate in a research survey. Women age 25 and above who are scheduled for an abdominal procedure and were seen in the General Surgery Clinic will be called and asked to complete a 5-10 minute verbal survey prior to their date of surgery. Some additional information will be gleaned from the medical record during the interview. Participation will be voluntary and all data collected will be recorded without any identifiers.

Part 2: A list of women 25 or older who are scheduled for an abdominal procedure after being seen in the General Surgery clinic will be generated to include MRN, procedure date, and pocedure type. A medical record review will be undertaken of these women and we will collect information about conditions that would facilitate or hinder the ability to perform a salpingectomy. No patient interaction will occur by the study team and all data will be de-identified at the time of collection. Data collected during this chart review will be linked and coded. Only coded data will be used during analysis. A separate password protected/encrypted file will contain the patient identifiers and the key to the coded sample numbers. This file will only be accessible by the PI or study team listed on this protocol on UVa premises, and will only be stored on a UVa server behind the UVa firewall, and will not be stored or accessed on personal computers. Thus, identified patient information will not be accessible to any individual, except the PI or study team listed on this protocol, ensuring protection of patient information

Study data will be analyzed to evaluate for acceptance of the program and acceptance of the mode of approaching the patient for counseling/consent. The frequency and types of conditions that hinder the ability to perform the suggested procedure will also be analyzed to determine how frequently the eligible population could receive a salpingectomy if a program was implemented.

ELIGIBILITY:
Inclusion Criteria:

* over 18 for Group 1
* over 25 for Group 2

Exclusion Criteria:

* male
* under 18 for Group 1
* under 25 for Group 2
* inability to give verbal consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Salpingectomy is a surgery only done on women.
Study Population: Women undergoing scheduled abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility and Acceptability from patients of opportunistic salpingectomy | 1 year
  based on responses to questionnaire , Likert scale of 1-5 with 1 low and 5 as high

IPD SHARING:
Plan to Share IPD: No